CLINICAL TRIAL: NCT06738303
Title: Carboplatin and Cabazitaxel Versus 177Lu-PSMA-617 in Patients With Aggressive, Metastatic Castrate-resistant Prostate Cancer (CATCH-177)
Brief Title: Cabazitaxel +/- Carboplatin vs 177Lu-PSMA-617 in Metastatic Castrate-resistant Prostate Cancer
Acronym: CATCH-177
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE13824
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Cabazitaxel; Lu-PSMA-617; Carboplatin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Carboplatin; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Cabazitaxel and carboplatin (Experimental): Cabazitaxel: Participants will receive cabazitaxel 20 mg/m2 as a one-hour intravenous infusion every three weeks for a total of 10 cycles or until disease progression, unacceptable toxicity.
  Carboplatin: Participants will receive carboplatin AUC 4 mg/mL/min every three weeks for a total of 10 cycles or until disease progression, unacceptable toxicity
  Interventions: Drug: Cabazitaxel and carboplatin
- Arm 2: Lu-PSMA-617 (Experimental): Participants will receive 177Lu-PSMA-617 7.4 GBq IV on Day 1 (+/-1 week) of each 6-week cycle for up to 6 cycles or until disease progression, unacceptable toxicity
  Interventions: Drug: Lu-PSMA-617

INTERVENTIONS:
Drug: Cabazitaxel and carboplatin — Given IV
  Arms: Arm 1: Cabazitaxel and carboplatin
Drug: Lu-PSMA-617 — Given IV
  Other Names: Pluvicto
  Arms: Arm 2: Lu-PSMA-617

SUMMARY:
The purpose of this study is to find out what treatment works best for participants with metastatic prostate cancer that are not responding to hormone treatment and docetaxel and are also Prostate-specific membrane antigen(PSMA) positive.

DETAILED DESCRIPTION:
Brief Background/Rationale

Metastatic prostate cancer initially is very responsive to androgen deprivation therapy (ADT), with intensification using an androgen receptor pathway inhibitor (ARPI) such as abiraterone acetate, enzalutamide, apalutamide, or darolutamide with or without docetaxel to prolong sensitivity to treatment and overall survival. Over time, however, prostate cancer transitions from castrate-sensitive to castrate-resistant. Metastatic castrate-resistant prostate cancer (mCRPC) has a dismal prognosis, with a median survival of under three years. There are now several agents with diverse mechanisms of action approved for use in mCRPC including cabazitaxel, sipuleucel-T, abiraterone acetate, enzalutamide, radium-223, olaparib, rucaparib, and 177Lu-PSMA-617.

Despite the treatment advances in the past decade, many cases of mCRPC either do not respond to these treatments or only respond for a short period of time. Predictive biomarkers are needed. In addition, with several options available, it is not always clear the optimal sequencing of these agents.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed metastatic castrate-resistant prostate cancer that has previously been treated with an androgen receptor pathway inhibitor. Prior docetaxel exposure is recommended but not mandatory. Tissue is not mandatory, but a pathologic report is required at time of enrollment.
2. Participants must have a PSMA-positive 18F-rhPSMA-7.3 performed within 12 weeks from C1D1 with ≥1 site with SUVmax ≥10) mCRPC with progression on prior novel hormonal agent to include at least one of the following:

   1. PSMA SUV mean <10
   2. ≥1 visceral metastasis
   3. ≥5 bone metastases

   OR two of the following
   1. TP53
   2. PTEN
   3. RB1 mutation.
3. Age > 18 years.
4. ECOG performance status of 0 to 2.
5. Subjects must have adequate organ and marrow function as defined below to be suitable for the randomized treatment outlined in this:

   * Absolute neutrophil count >1000/μL; platelet count >90 000/μL; hemoglobin >8.5 g/dL) at screening.

   Note: Subjects must not have received any growth factors within 7 days or blood transfusions within 14 days prior to the hematologic laboratory values obtained at screening).
   * Total bilirubin (TBIL) <2.5 × the upper limit of normal (ULN) at screening, except subjects with documented Gilbert syndrome who must have a TBIL <3 mg/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 ULN at screening
   * Creatinine clearance ≥40 mL/min and/or estimated glomerular filtration rate (eGFR) ≥30
   * Albumin >30 g/L (3.0 g/dL) at screening
6. Subjects receiving bisphosphonates or other approved bone-targeting therapy (e.g., denosumab) must be on a stable dose for at least 14 days before the start of study treatment.
7. Subjects of child-producing potential agree to use highly effective contraceptive methods (i.e., barrier contraception measures such as a male condom with spermicide during intercourse) and avoid sperm donation during the study treatment and for 3 months after the last dose of study treatment. A man is considered to be of child producing potential, unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy. Partners of participants must also practice approved forms of birth control
8. Subjects must have the ability to understand and the willingness to sign a written informed consent form (ICF).
9. Members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Evidence of hormone-sensitive prostate cancer (HSPC)
2. Evidence of small cell prostate cancer
3. Subjects receiving any other investigational agents.
4. Diagnosis of another clinically significant malignancy within the previous 2 years other than curatively treated non-melanomatous skin cancer or superficial urothelial carcinoma and other in situ or noninvasive malignancies, as determined by the PI or Co-PI.
5. Subjects with brain metastases/central nervous system (CNS) disease that are treated prior to enrollment will be allowed in this clinical trial.
6. Known or suspected significant hypersensitivity to any components of the formulation used for Cabazitaxel, carboplatin or 177Lu-PSMA-617.
7. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations considered by the Investigator to limit compliance with study requirements.
8. Prior treatment toxicities not resolved to ≤ Grade 2 according to NCI CTCAE Version 5.0

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PSA response rate as assessed by the change in PSA ratio | Baseline, 12 weeks post intervention
  PSA decline of ≥50% (PSA50) at 12 weeks. PSA decline will be measured by obtaining the ratio of PSA obtained on cycle 5 day 1 to baseline PSA obtained cycle 1 day 1.

SECONDARY OUTCOMES:
Progression Free Survival | Upto 26 weeks
Time to next systemic therapy | Cycle 1 day1(each cycle will be 6 weeks upto 10 cycles) to the first day of subsequent systemic cancer-directed therapy

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Barata, MD, MSc, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code